CLINICAL TRIAL: NCT00908141
Title: Immunologic Effects of GM-CSF (Sargramostim, Leukine®) in Patients With Biochemically-relapsed Prostate Cancer
Brief Title: GM-CSF in Treating Patients With Relapsed Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE6805; P30CA043703 (NIH); CASE6805 (Other: Case Comprehensive Cancer Center); 8201 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: sargramostim (days1-14) (Experimental): Patients receive sargramostim (GM-CSF) subcutaneously (SC) on days 1-14. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: sargramostim
- Arm II: sargramostim (3xweek) (Experimental): Patients receive GM-CSF SC three times weekly for 4 weeks. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: sargramostim

INTERVENTIONS:
Biological: sargramostim — Given subcutaneously on varying schedule

SUMMARY:
RATIONALE: Colony stimulating factors, such as GM CSF, may increase the number of immune cells found in bone marrow or peripheral blood. It is not yet known which GM-CSF regimen is more effective in treating patients with prostate cancer.

PURPOSE: This randomized phase II trial is studying how well GM-CSF works in treating patients with relapsed prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the ability of sargramostim (GM-CSF) to increase the number and activation of dendritic cells (DC) in patients with biochemically relapsed prostate cancer.

Secondary

* To determine the effect of administration schedule and hormonal state on sargramostim-induced DC number and activation in these patients.
* To correlate the effects of sargramostim on DC number and activation with effects on prostate-specific antigen (PSA) modulation.
* To determine whether sargramostim administration generates antiprostate cancer immune responses in these patients.

OUTLINE: Patients are stratified according to hormonal status (androgen-dependent vs androgen-independent). Patients are then randomized to 1 of 2 treatment arms.

* Arm I: Patients receive sargramostim (GM-CSF) subcutaneously (SC) on days 1-14. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive GM-CSF SC three times weekly for 4 weeks. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for dendritic cell (DC) number by flow cytometry, DC activation by quantitative real-time polymerase chain reaction (QRT-PCR), and immunity by serological analysis of recombinant cDNA expression libraries (SEREX).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Non-metastatic, recurrent systemic disease as manifested by a rising PSA, defined as ≥ 2 consecutive rises in PSA to be documented over a reference value (measure 1)

    * The first rising PSA (measure 2) should be at taken ≥ 14 days after the reference value
    * A third confirmatory PSA measure is required (second beyond the reference level) to be greater than the second, and it must be obtained ≥ 14 days after the second measure

      * If this is not the case, a fourth PSA is required to be taken and be greater than the second measure
    * No local-only relapse
* Must have undergone prior definitive therapy for prostate cancer consisting of external beam radiotherapy, brachytherapy (with or without external beam radiotherapy), or radical prostatectomy (with or without adjuvant androgen ablation)

  * Patients who have not undergone definitive therapy as above or who have undergone hormonal therapy alone are not eligible
* No evidence of metastases on bone or CT scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Leukocytes ≥ 3,000/μl
* Absolute neutrophil count ≥ 1,500/μl
* Platelets ≥ 100,000/μl
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* No active thrombophlebitis or disseminated intravascular coagulopathy
* No history of pulmonary embolus
* No history of immunodeficiency or autoimmune diseases
* No uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy for any reason
* No concurrent anticoagulation therapy (i.e., therapeutic coumadin)

  * Prophylactic anticoagulation (e.g., aspirin) allowed
* No concurrent systemic corticosteroids or other immunosuppressives

  * Inhaled or topical steroids allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, MD, FACP, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from local medical clinic from June 2006 to August 2010.
Groups:
- Group A: Sargramostim (Days 1-14): GROUP A:
  Sargramostim 250ug/m2/day subcutaneously (s.c.) on days 1-14 of a 28-day cycle
- Group B:Sargramostim (3 x Week): GROUP B:
  Sargramostim 250ug subcutaneously (s.c.) three times a week continuously
Period: Overall Study
Arm/Group | Group A: Sargramostim (Days 1-14) | Group B:Sargramostim (3 x Week)
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group B: Sargramostim (3 x Week): GROUP B:
  Sargramostim 250ug subcutaneously (s.c.) three times a week continuously
- Total: Total of all reporting groups
Arm/Group | Group A: Sargramostim (Days 1-14) | Group B: Sargramostim (3 x Week) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Customized [Number; unit: participants]
  40-49 years | 1 | 0 | 1
  50-59 years | 2 | 2 | 4
  60-69 years | 2 | 4 | 6
  70-79 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response
Description: The number of patients with PSA modulation defined as PSA decline of at least 50%
Time Frame: post treatment at 9 weeks
Measure: Number; unit: participants
Arm/Group | Group A: Sargramostim (Days 1-14) | Group B: Sargramostim (3 x Week)
Number analyzed (Participants) | 8 | 8
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: All patients will be evaluable for toxicity from the time of their first treatment with sargramostim through follow up over an approximate three year period.
Arm/Group | Group A: Sargramostim (Days 1-14) | Group B: Sargramostim (3 x Week)
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Sargramostim (Days 1-14) (N=8) | Group B: Sargramostim (3 x Week) (N=9)
Thrombosis (Vascular disorders) | 0 | 1
Ureteral obstruction (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Sargramostim (Days 1-14) (N=8) | Group B: Sargramostim (3 x Week) (N=9)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine, elevated (Investigations) | 0 | 2
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1 | 0
Elevated SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 0 | 1
Elevated SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 0 | 1
Fatigue (General disorders) | 3 | 2
Flu-like Symptoms (General disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 1 | 0
GI symptoms of nausea, emesis, and diarrhea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemoglobin (Investigations) | 1 | 2
Hemoglobinuria (Renal and urinary disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Infection with normal ANC, intermittent (Blood and lymphatic system disorders) | 0 | 1
Infection with unknown ANC(Absolute neutrophil count) (Blood and lymphatic system disorders) | 0 | 1
Injection site reaction (Skin and subcutaneous tissue disorders) | 7 | 8
Insomnia (Psychiatric disorders) | 1 | 0
Intermittent rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Mid-low back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgias (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 1
Pain (Back and Left arm) (General disorders) | 1 | 0
Pain Left buttock (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, Right knee (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, sciatic (right) (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes